CLINICAL TRIAL: NCT03067753
Title: Monosialoganglioside Ganglioside in Cerebral Radiation Necrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2016-HN02
Record Dates: First submitted 2017-01-10; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Cerebral Radiation Necrosis
MeSH Terms: interventions — G(M1) Ganglioside; Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed steroid (Active Comparator): Pulse steroid, methylprednisolone, was administered by intravenous infusion over 3 consecutive days. Three grams of methylprednisolone was given in each cycle. Administration of 1 g was infused over 1 h daily for 3 days on an in-patient basis, which then tailed off in 10 days with administration of oral prednisolone.
  Interventions: Drug: Methylprednisolone (Steroid Hormone); Drug: Prednisolone
- Monosialoganglioside ganglioside (Experimental): Monosialoganglioside ganglioside was given at 100 mg/time, once a day for 2 months.
  Interventions: Drug: Monosialoganglioside Ganglioside

INTERVENTIONS:
Drug: Monosialoganglioside Ganglioside — Monosialoganglioside ganglioside was given at 100 mg/time, once a day for 2 months.
  Arms: Monosialoganglioside ganglioside
Drug: Methylprednisolone (Steroid Hormone) — Pulse steroid, methylprednisolone, was administered by intravenous infusion over 3 consecutive days. Three grams of methylprednisolone was given in each cycle. Administration of 1 g was infused over 1 h daily for 3 days on an in-patient basis, which then tailed off in 10 days with administration of oral prednisolone.
  Arms: Pulsed steroid
Drug: Prednisolone
  Arms: Pulsed steroid

SUMMARY:
Monosialoganglioside Ganglioside in Cerebral Radiation Necrosis

DETAILED DESCRIPTION:
A prospective phase II trial was conducted to test the efficacy of monosialoganglioside ganglioside for the treatment of cerebral radiation necrosis

ELIGIBILITY:
Inclusion Criteria:

* Undergone only one course of definitive radiotherapy for histologically confirmed nasopharyngeal carcinoma years before;
* At least two consecutive MRI study supporting the diagnosis of cerebral radiation necrosis(CRN) with an interval of 3-4 months, with the second MRI showing progressive disease compared with the first MRI;
* Progressive neurologic symptoms or signs;
* Mini-mental status examination(MMSE) score must be ≤27;
* Karnofsky performance status≥70 ;
* Supposed to live more than 6 months.

Exclusion Criteria:

* After the second course of radiotherapy for recurrent nasopharyngeal carcinoma;
* Local or regional relapse,or with distant metastasis;
* Cerebrovascular disease;
* Second primary malignancy;
* Diabetes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From the first day of treatment, to 3 months after treatment
  Response Evaluation Criteria in Solid Tumors (RECIST) were used.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No